CLINICAL TRIAL: NCT02505516
Title: BLADDER CANCER SCREENING AMONG DIABETIC PATIENTS ON METFORMIN THERAPY IN A WEST AFRICA SUB-REGION
Brief Title: BLADDER CANCER SCREENING AMONG DIABETIC PATIENTS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UFUOMA MILLER FAKPOR (Other)
Responsible Party: Sponsor-Investigator, UFUOMA MILLER FAKPOR, miss, University of Cape Coast
Organization: University of Cape Coast (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 021
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Bladder Cancer; Diabetes
Keywords: pathology
MeSH Terms: conditions — Urinary Bladder Neoplasms; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Placebo Comparator): metformin 500mg
  Interventions: Other: metformin
- not on metformin (No Intervention)

INTERVENTIONS:
Other: metformin
  Other Names: glucophage
  Arms: metformin

SUMMARY:
patients om metformin from diabetic clinic were checked for bladder cancer

ELIGIBILITY:
Inclusion Criteria:

* 150 people attending diabetic clinic

Exclusion Criteria:

Ages: 25 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of diabetic patients on metformin therapy | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universty of Capecoast, Cape Coast, Ghana